CLINICAL TRIAL: NCT00770939
Title: A Cohort Study to Evaluate the Effect of Vivostat Platelet Rich Fibrin on Diabetic Foot Ulcers.
Brief Title: Evaluation of the Effect of Vivostat Platelet Rich Fibrin(PRF) in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vivostat (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-001
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Diabetic Foot Ulcers
Keywords: Complete healing of chronic diabetic foot ulcers; Platelet Rich Fibrin; Vivostat; Growth factor treatment; Treatment of chronic diabetic foot ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vivostat PRF — Ulcer will be treated week 1,2,3,4,5 and 6 with Vivostat PRF

SUMMARY:
Diabetic foot ulcers are a challenge to health care professionals because there are only few effective topical therapeutic interventions.

Growth factor treatment has shown to be beneficial for healing of diabetic foot ulcers in conjunction with extensive surgical debridement. Autologues platelet releasate which contains platelet derived growth factor appears to be more effective than standard therapy in case studies.

This protocol will evaluate the healing effect of Vivostat PRF treatment of non-eschemic foot ulcers to identify responders and to enable sample size calculation for a subsequent pivotal trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 weeks history (with wound area measurements) within a wound care institution before the first visit (week -3). In case of referral the patient history must be documented
* All patients must complete a 3 week screening period i.e. they will be interviewed and accessed at the first meeting. During the 3 week period patient compliance will be monitored.
* Age >18 years
* Type I or Type II Diabetes Mellitus
* Ulcer at or below the ankle which has been present for at least 4 weeks, and has received best practice care
* Ulcer area between 0,5 and 16 cm2
* If there is more than one ulcer or bilateral ulcers, the investigator shall choose the one index ulcer to be treated (typically the largest one). The other ulcers will receive standard care and is not included in the study
* Ulcer type: University of Texas grade IA.
* Evidence of adequate arterial perfusion: Toe pressure reading of ≥ 30 mmHg or if toe is missing, transcutaneous oxygen (TcPO2) of ≥ 30mmHg on the foot.
* Patient foot is appropriately off loaded (contact cast, pneumatic walking cast)
* Orthopaedic assessment has been completed to rule out a mechanical source of ulceration
* Relative wound area reduction less than 50% from week -3 to week 0 (pre-screening period)
* Signed informed consent

Exclusion Criteria:

* Clear indication for surgery (vascular reconstruction or skin transplant)
* Ulcer with exposed bone or tendon
* Bone involvement (probe to bone or x-ray)
* Patients with 3 ulcers or more at the foot investigated
* Osteomyelitis
* Clinical signs of infections
* Necrosis in the wound (one week into the screening period).
* Patients with known MRSA
* Malnutrition. Albumin < 2,5g/dl
* Ulcers resulting from electrical, chemical, radiation burns
* HbA1c > 12%
* Male: Hb < 8 mmol/l (12,9 g/dlFemale: Hb < 7 mmol/l (11,3 g/dl)
* Platelet count <140 *109/l
* Pregnancy and fertile women not practicing sufficient birth control
* Fertile women having a positive pregnancy test week 0 Lactating women
* Patients on haemodialysis
* History of peripheral vascular repair within 4 weeks prior to study enrollment
* Bleeding disorders, haemophilia, sickle cell disease, thrombocytopenia, and leukaemia or blood dyscrasias
* Current treatment for malignancy or neoplastic disease or collagen vascular disease
* Highly communicable disease or diseases that may limit follow - up (e.g. immunocompromised conditions, hepatitis, active tuberculosis)
* Patient has inadequate venous access to draw blood
* History of alcohol or drug abuse within the last year prior to randomization
* Patient known to have psychological, developmental, physical, emotional or social dis-order or other ailments that may interfere with the study requirements
* Patients enrolled in an other clinical trial for wound treatment within 30 days prior to enrollment
* Non-compliance in the screening period
* Patients who have received growth factor therapy e.g. becaplermin within 7 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Proportion of completely healed ulcers after 12 weeks | 12 weeks
Percentage of patients with a 50% reduction of wound area after 4 and 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Granulation rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ruge, Study Director — Vivostat
Locations (5):
- Woundhealing Centre Bispebjerg Hospital, Copenhagen, Denmark
- Germany (3):
  - Diabetes Klinik Bad Mergentheim GmbH, Bad Mergentheim
  - Gesundheitszentrum Mathias Hospital, Rheine
  - Krankenhaus der Barmherzigen Brüder, Trier
- Diabetes/ Endokrin sektion, Lund, Sweden